CLINICAL TRIAL: NCT04241003
Title: Effects of the SmartDrive on Mobility, Activity and Shoulder Pain Among People With SCI Using Manual Wheelchairs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Permobil, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Per2018M01
Record Dates: First submitted 2020-01-16; First posted 2020-01-27 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2021-01

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- SmartDrive - baseline and intervention (Experimental): One arm for all users. Baseline - two weeks data collection documenting usage of wheelchair prior to intervention. Introduction of SmartDrive, a time period to get used to the SmartDrive and then two weeks data collection documenting usage of wheelchair with the intervention.
  Interventions: Device: SmartDrive Mx2+

INTERVENTIONS:
Device: SmartDrive Mx2+ — Rear-mounted power assist

SUMMARY:
This is a prospective study of manual wheelchair users with spinal cord injury (SCI). The users will be their own controls. The primary purpose of the study is to evaluate the ability of the power assist device SmartDrive to increase the ability to be mobile.

DETAILED DESCRIPTION:
The hypothesis of the study is that the SmartDrive will enable the user to be more active, both in commuting longer distances with less strokes needed, and managing single difficulties stopping them from activity. The two assessments selected, distance travelled and the daily diary, should directly reflect the impact of the SmartDrive. In addition, the the International Spinal Cord Society (ISCoS) pain data set, Wheelchair User's Shoulder Pain Index (WUSPI) and Wheelchair Outcome Measure (WhOM) will be used. In WhOM, the participants will state some activities they perform in their wheelchair that are important to them, and how satisfied they are with their current level of performance of that activity. After the intervention period the satisfaction is reassessed. This will enable to capture the effect SmartDrive usage has on the participant's daily life (beyond distance commuted and pain level).

After enrollment, the participants will be followed for two weeks using their wheelchair without SmartDrive. After attaching the SmartDrive, they will have three weeks to get into a use of the device on a regular basis in their everyday life, and then follows two consecutive weeks of study intervention and data collection. To capture the long-term effect and allow for season variability, follow-up data will be collected at three and six months after start of study intervention.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent which includes compliance with the requirements listed in the informed consent form (ICF) and in this protocol
* 18 years of age inclusive, at the time of signing the informed consent.
* Motor level C6-L3 Spinal Cord Injury, American Spinal Injury Association Impairment Scale (AIS) A-C since at least six months
* Full time manual wheelchair users, able to propel their own wheelchairs independently
* Eligible reason for SmartDrive prescription (Self-reported shoulder pain, and/or decreased physical endurance for propulsion, limiting user from activity)

Exclusion Criteria:

* Cognitive impairment affecting the ability to operate the SmartDrive, as deemed by prescribing clinician
* Weigh more than 150 kilos due to the technical specification of the SmartDrive
* Currently participating in another clinical study anticipated to affect the outcome or ability to compete this study
* Planned change from daily routines during the following two months, such as holiday, move, change jobs
* For any other reason not suitable for participation in the study, as deemed by prescribing clinician
* Do not use a smart phone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-06-11 (Actual); Primary Completion 2020-11-09 (Actual); Study Completion 2021-05-14 (Actual)

PRIMARY OUTCOMES:
Change in wheelchair usage per day (time) | Two weeks during baseline (without SmartDrive) and two weeks during intervention (with SmartDrive)
  Data captured by study specific smart watch to document usage of wheelchair
Change in wheelchair usage per day (distance) | Two weeks during baseline (without SmartDrive) and two weeks during intervention (with SmartDrive)
  Data captured by study specific smart watch to document usage of wheelchair
Change in activity level of patient reported wheelchair use | Two weeks during baseline (without SmartDrive) and two weeks during intervention (with SmartDrive)
  Paper diary for activity level (high, medium, low) rated by the participant every evening.

SECONDARY OUTCOMES:
Pain in upper extremities, WUSPI | At visit 2 and 3 (start and end of intervention) and at 3 and 6 months Follow up for a period of up to one year
  Wheelchair user shoulder pain index (WUSPI). WUSPI is a simple and effective self-report questionnaire for quickly measuring the functional cost of shoulder pain in wheelchair users. The WUSPI targets activity limitation resulting from shoulder pain (4 subsections), including wheelchair transfers, wheelchair mobility, selfcare and general activities.
Pain in upper extremities, ISCOS | At visit 2 and 3 (start and end of intervention) and at 3 and 6 months Follow up for a period of up to one year
  The International Spinal Cord Injury Pain Basic Data Set is a questionnaire addressing clinically relevant core questions concerning SCI-related pain.
Wheelchair Outcome Measure WhOM | At visit 2 and 3 (start and end of intervention) and at 3 and 6 months Follow up for a period of up to one year
  The WhOM is a client-centred two-part measure of wheelchair and seating system intervention, documenting expectations of the new intervention (part 1) which is followed up in the second part.
Change in pain level of patient reported wheelchair use | Two weeks during baseline (without SmartDrive) and two weeks during intervention (with SmartDrive)
  Paper diary for pain score on a Likert scale rated by the participant every evening.

CONTACTS AND LOCATIONS:
Overall Officials: Claes Hultling, Prof., Principal Investigator — Spinalis
Locations (1):
- Stiftelsen Spinalis, Solna, Sweden

IPD SHARING:
Plan to Share IPD: No